CLINICAL TRIAL: NCT06024109
Title: Prospective, International, Randomized, Multicentric, Controlled Study on the Performance of SYMMCORA® Mid-term Unidirectional Barbed Suture Versus V-loc® Suture Material in Patients Undergoing Laparoscopic Total Hysterectomy
Brief Title: Performance of SYMMCORA® vs. V-Loc® Suture Material in Patients Undergoing Laparoscopic Total Hysterectomy
Acronym: BARHYSTER
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2001
Record Dates: First submitted 2023-08-15; First posted 2023-09-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Abnormal Uterine Bleeding; Endometriosis; Uterine Prolapse; Uterine Cancer; Ovarian Cancer; Fallopian Tube Cancer; Cervical Cancer; Endometrial Cancer
Keywords: Barbed Suture; Hysterectomy; Laparoscopy; Minimal Invasive
MeSH Terms: conditions — Metrorrhagia; Endometriosis; Uterine Prolapse; Uterine Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Sutures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SYMMCORA®: Barbed suture SYMMCORA® used for the vaginal cuff closure in female patients undergoing total laparoscopic hysterectomy. The product under investigation and the comparator suture material will be used in routine clinical practice and according to the Instructions for Use (IfU).
  Interventions: Device: Closure of the Vaginal Cuff after Total Hysterectomy
- V-Loc®: Barbed suture V-Loc® used for the vaginal cuff closure in female patients undergoing total laparoscopic hysterectomy. The product under investigation and the comparator suture material will be used in routine clinical practice and according to the Instructions for Use (IfU).
  Interventions: Device: Closure of the Vaginal Cuff after Total Hysterectomy

INTERVENTIONS:
Device: Closure of the Vaginal Cuff after Total Hysterectomy — Closure of the vaginal cuff in patients undergoing laparoscopic total hysterectomy. The product under investigation and the comparator suture material will be used in routine clinical practice and according to the Instructions for Use (IfU).
  Other Names: Suturing

SUMMARY:
The aim of this study is to show the superiority of the new unidirectional barbed suture (SYMMCORA® mid-term, unidirectional) to conventional suture material in terms of time to perform the vaginal cuff closure during gynecologic surgeries without an increase in the complication rate.

Secondly, the superiority of SYMMCORA®, mid-term unidirectional compared to the V-Loc®, unidirectional will be assessed regarding the mean time to close the vaginal cuff. The study will be performed in routine clinical setting, the only difference will be the randomization into two different suture groups. Both suture materials which will be applied to approximate the vaginal cuff are approved and carrying the CE-marks. Additionally, both sutures will be applied in their intended use. Neither additional invasive measures nor additional burden in regard to the patient will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing an elective, laparoscopic total hysterectomy
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Open surgery
* Patients undergone immunosuppressive drug treatment within the prior 6 months
* Patients with hypersensitivity or allergy to the suture material.
* Participation in another clinical study
* Non-compliance of patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing an elective, laparoscopic total hysterectomy
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Suturing time to close the vaginal cuff | intraoperatively
  Measured in Minutes. Time to perform the vaginal cuff closure after laparoscopic total hysterectomy using a stop watch. Time starts when the needle passes the first time the tissue and ends after completion of the wound closure (cut of the needle from the thread).

SECONDARY OUTCOMES:
Number of patients with early complications | at discharge (up to 10 days after surgery)
  Documented early complications include Hemoglobin drop and Fever more than 38°C within 48 hours
Number of patients with complications over the study period | at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  Documented complications include Vaginal cuff infection, Vaginal cuff dehiscence (Defined as a visually confirmed partial or complete opening of the vaginal stump with or without visceral organ herniation), Vaginal cuff granulation formation, Pelvic Abscess Formation, Hematoma, Vaginal spotting (defined as bloody vaginal discharge that did not require extraordinary procedures or medication and disappeared spontaneously. (Days of postoperative bleeding, Number of pads / tampons used), Vaginal bleeding (Defined as postoperative vaginal stump bleeding that required additional stump suture to stop bleeding. (Days of postoperative bleeding, number of pads / tampons used), Urinary tract infection, Bladder injury, Ureter injury, Bowel obstruction, Ileus, Cystitis and Pelvic Adhesions.
Number of patients with device deficiencies over the study period | intraoperatively, at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  Documented device deficiencies include Suture rupture, Knots in the thread, Connection between needle and thread not intact and Disconnection of the anchor from the thread
Patient satisfaction (VAS 0-100) over time | at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  The patient's self assessment of her satisfaction with the surgery. This parameter will be noted using the Visual Analogue Scale (VAS), represented by a line 10 cm of length, which states "0" at one end representing "low" and "100" at the opposite end representing "high". The value is measured in [mm] with a ruler and documented in whole numbers.
Progress of Female Sexual Function Index (FSFI) compared to baseline | Preoperatively (baseline), at follow-up visits 6-8 weeks postoperatively and 6 months postoperatively
  The Female Sexual Function Index (FSFI) is a 19-item, self-report measure of female sexual function that provides scores on overall levels of sexual function as well as the primary components of sexual function in women, including sexual desire, arousal, orgasm, pain, and satisfaction. The 19 items of the FSFI use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning on the respective item. (0 points in some cases for items that are not applicable). To score the measure, the sum of each domain score is first multiplied by a domain factor ratio (0.6 for desire; 0.3 for arousal and lubrication; 0.4 for orgasm, satisfaction and pain) in order to place all domain totals on a more comparable scale, and then subsequently summed to derive a total FSFI score. The domain scores range from 1.2 - 6, the overall score ranges from 7.2 - 36.
Overall operation time | intraoperatively
  From the first cut to the end of the surgery
Cost of treatment | at discharge (approximately 10 days after surgery)
  Calculation using the length of hospitalization (days until discharge), suturing time, suture costs and needed transfusions)
Length of postoperative hospital stay | at discharge (approximately 10 days after surgery)
  calculated by subtracting the surgery date from the date of discharge
Progress of Patient's abdominal pain (VAS 0-100) compared to baseline | preoperatively (baseline) and at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  The patient's self assessment of her abdominal pain. This parameter will be noted using the Visual Analogue Scale (VAS), represented by a line 10 cm of length, which states "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain". The value is measured in [mm] with a ruler and documented in whole numbers
Progress of Patient's pelvic pain (VAS 0-100) compared to baseline | preoperatively (baseline) and at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  The patient's self assessment of her pelvic pain. This parameter will be noted using the Visual Analogue Scale (VAS), represented by a line 10 cm of length, which states "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain". The value is measured in [mm] with a ruler and documented in whole numbers
Progress of Patient's lumbar pain (VAS 0-100) compared to baseline | preoperatively (baseline) and at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  The patient's self assessment of her lumbar pain. This parameter will be noted using the Visual Analogue Scale (VAS), represented by a line 10 cm of length, which states "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain". The value is measured in [mm] with a ruler and documented in whole numbers
Progress of General Health Status compared to baseline | preoperatively (baseline) and at discharge (up to 10 days after surgery), 6-8 weeks postoperatively, 6 months postoperatively
  The patient's self assessment of her general health status. Health status is based on assessment of the patient to the question, "Would you say your health in general is...:" The options are excellent / very good / good / fair / poor
Patient assessment of postoperative Dyspareunia | at both follow-up visits (6-8 weeks postoperatively and 6 months postoperatively)
  Dyspareunia is defined by genital pain that can be experienced before, during, or after intercourse. The patient answers with yes or no.
Assessment of the handling of the barbed suture (SYMMCORA®) | intraoperatively
  Assessment of the handling of the unidirectional barbed suture (SYMMCORA®) intra-operatively including eleven different dimensions (pliability, Pass-through, traumaticity, anchoring capacity, safety of closure, locking system size, locking system deployment, locking system unbarbed area, locking system safety of closure, atraumaticity, wound closure approximation) and an overall impression with 5 evaluations levels (excellent, very good, good, satisfied, poor).
Assessment of the handling of the barbed suture (SYMMCORA®) compared to conventional suture | intraoperatively
  Assessment of the handling of the barbed suture (SYMMCORA®) compared to conventional suture regarding degree of difficulties and the ease of handling. (Likert Scale: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree).
Assessment of the handling of the barbed suture (SYMMCORA®) compared to barbed suture (V-Loc) | intraoperatively
  Assessment of the barbed suture (SYMMCORA®) compared to barbed suture (V-Loc®) regarding smoothness, suppleness, traumaticity of the thread, the handling, the opening of the package and the overall opinion (Likert Scale: worse, equal, better).

CONTACTS AND LOCATIONS:
Overall Officials: Amadeus Hornemann, Prof. Dr., Principal Investigator — Klinikum Sachsenhausen der DGD
Locations (2):
- Klinikum Sachsenhausen der DGD, Frankfurt am Main, Hesse, Germany
- Hospital Sant Joan de Déu de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumann P, Sanchez LH, Garcia NG, Sologiuc L, Hornemann A. Assessment of a novel unidirectional mid-term absorbable barbed suture versus a competitor barbed suture for vaginal cuff closure after gynaecology surgery, study protocol of a randomized controlled trial - BARHYSTER. BMC Surg. 2025 Jan 14;25(1):23. doi: 10.1186/s12893-024-02700-z. PMID 39806425